CLINICAL TRIAL: NCT00800540
Title: Effects of Topical Hypotensive Drugs on Circadian Ocular Perfusion Pressure and Ocular Blood Flow in Patients With Open-Angle Glaucoma
Brief Title: Circadian Ocular Perfusion Pressure and Ocular Blood Flow
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: C-07-16; 2007-005936-99 (EudraCT Number)
Record Dates: First submitted 2008-12-01; First posted 2008-12-02 (Estimated); Results first posted 2013-03-22 (Estimated); Last update posted 2013-03-22 (Estimated); Status verified 2013-03

CONDITIONS: Glaucoma
Keywords: glaucoma; ocular perfusion pressure; ocular blood flow; open angle glaucoma requiring more than one IOP-lowering medication
MeSH Terms: conditions — Glaucoma | interventions — brinzolamide; Timolol; Azarga; Brimonidine Tartrate; Ophthalmic Solutions; Brimonidine Tartrate, Timolol Maleate Drug Combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- AZARGA/COMBIGAN (Other): AZARGA, followed by COMBIGAN, as randomized. Each fixed combination instilled in the study eye, one drop twice daily (9:00 and 21:00), for six weeks, with a 4-week washout period separating the two treatment periods.
  Interventions: Drug: Brinzolamide 10 mg/ml/Timolol 5 mg/ml eye drops suspension; Drug: Brimonidine 20 mg/ml/Timolol 5 mg/ml eye drops solution
- COMBIGAN/AZARGA (Other): COMBIGAN, followed by AZARGA, as randomized. Each fixed combination instilled in the study eye, one drop twice daily (9:00 and 21:00), for six weeks, with a 4-week washout period separating the two treatment periods.
  Interventions: Drug: Brinzolamide 10 mg/ml/Timolol 5 mg/ml eye drops suspension; Drug: Brimonidine 20 mg/ml/Timolol 5 mg/ml eye drops solution

INTERVENTIONS:
Drug: Brinzolamide 10 mg/ml/Timolol 5 mg/ml eye drops suspension — Fixed combination ophthalmic suspension
  Other Names: AZARGA™
Drug: Brimonidine 20 mg/ml/Timolol 5 mg/ml eye drops solution — Fixed combination ophthalmic solution
  Other Names: COMBIGAN®

SUMMARY:
The purpose of this study was to compare the short term effects of two intraocular pressure (IOP) lowering medications on ocular perfusion pressure (OPP), ocular blood flow, intraocular pressure, and blood pressure in patients with glaucoma. Ocular perfusion pressure (OPP) is defined as the difference between arterial blood pressure (diastolic and systolic) and intraocular pressure. The primary efficacy assessment is based on diastolic ocular perfusion pressure.

ELIGIBILITY:
Inclusion Criteria:

* Sign Informed Consent.
* Diagnosis of open-angle glaucoma in at least one eye.
* Requires more than one IOP-lowering medication.
* IOP measurements at Screening, Safety, and Eligibility/Period 1 Baseline Visits as specified in protocol.
* Able to discontinue all IOP-lowering medication prior to Eligibility Visit and for 4 weeks between treatment periods.
* Willing to complete all required study visits.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Female of child-bearing potential if pregnant, lactating, or not using highly effective birth control measures.
* Severe central visual field loss in either eye.
* Previous glaucoma surgery in the study eye.
* Intraocular surgery in the study eye within 3 months prior to the Screening Visit.
* Wears contact lenses.
* Allergy/hypersensitivity to study medication.
* Cannot safely discontinue use of glucocorticoid medication.
* Uses medication that could affect IOP or blood pressure.
* Recent use of high-dose aspirin.
* Bronchial asthma or severe chronic obstructive pulmonary disease.
* Diabetic retinopathy.
* Any abnormality preventing reliable tonometry.
* Any severe illness or condition unsuitable for the study, in the opinion of the investigator.
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2009-02; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Contact Alcon Call Center at 1-888-451-3937 For Trial Locations, Fort Worth, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from and enrolled at one study center located in Greece.
Groups:
- AZARGA/COMBIGAN: AZARGA, followed by COMBIGAN, as randomized. Each fixed combination was used for 6 weeks, with a 4-week washout period separating the two treatment periods.
- COMBIGAN/AZARGA: COMBIGAN, followed by AZARGA, as randomized. Each fixed combination was used for 6 weeks, with a 4-week washout period separating the two treatment periods.
Period: Period One: 6 Weeks
Arm/Group | AZARGA/COMBIGAN | COMBIGAN/AZARGA
Started | 17 | 18
Completed | 16 | 17
Not Completed | 1 | 1
Not completed — Noncompliance | 1 | 0
Not completed — Pt Decision Unrelated to Adverse Event | 0 | 1
Period: Washout: 4 Weeks
Arm/Group | AZARGA/COMBIGAN | COMBIGAN/AZARGA
Started | 16 | 17
Completed | 16 | 17
Not Completed | 0 | 0
Period: Period 2: 6 Weeks
Arm/Group | AZARGA/COMBIGAN | COMBIGAN/AZARGA
Started | 16 | 17
Completed | 16 | 16
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Population: This reporting group includes all enrolled participants.
Groups:
- Overall: All enrolled
Arm/Group | Overall
Number analyzed (Participants) | 35
Age Continuous [Mean (Standard Deviation); unit: years] | 65.2 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 16
Region of Enrollment [Number; unit: participants]
  Greece | 35

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Overall Diastolic Ocular Perfusion Pressure at Week 6
Description: Diastolic ocular perfusion pressure (DOPP) is defined as the difference between diastolic arterial pressure and intraocular pressure. Diastolic arterial pressure was measured with a calibrated automated sphygmomanometer. Intraocular pressure was measured with a calibrated pneumatonometer. A lower DOPP indicates a lower optic blood supply, which can be a risk factor for developing glaucoma or glaucoma progression (leading to optic nerve damage).
Time Frame: Week 0, Week 6 (period-based)
Population: This reporting group includes all patients who received study medication and completed the on-therapy follow-up study visit in both periods (ITT).
Measure: Mean (Standard Error); unit: mmHg (millimeters of mercury)
Units Other Than Participants: eyes
Groups:
- AZARGA; COMBIGAN: One drop in the study eye, twice daily (9:00 and 21:00), for six weeks
Arm/Group | AZARGA | COMBIGAN
Number analyzed (Participants) | 32 | 32
Number analyzed (eyes) | 41 | 41
mmHg (millimeters of mercury) | 2.6 (0.780) | 0.8 (0.779)

2. Secondary Outcome: Mean Change From Baseline in Circadian Diastolic Ocular Perfusion Pressure at Week 6
Description: Circadian diastolic ocular perfusion pressure (COPP) is defined as the variations in diastolic OPP during the day and night. Diastolic ocular perfusion pressure was calculated at 7 timepoints over a 24-hour period. Changes in the diastolic ocular perfusion pressure rhythm throughout the day (outside the normal range) may affect glaucoma progression.
Time Frame: Week 0, Week 6 (period-based)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: mmHg (millimeters of mercury)
Units Other Than Participants: eyes
Arm/Group | AZARGA | COMBIGAN
Number analyzed (Participants) | 32 | 32
Number analyzed (eyes) | 41 | 41
mmHg (millimeters of mercury)
  9:00 am | 2.8 (1.282) | 6.5 (1.282)
  1:00 pm | 3.0 (1.282) | 2.1 (1.282)
  5:00 pm | 4.4 (1.282) | 3.9 (1.282)
  9:00 pm | 4.5 (1.282) | 2.0 (1.282)
  12:00 am | 0.8 (1.282) | -5.6 (1.282)
  3:00 am | 0.3 (1.282) | -4.0 (1.282)
  6:00 am | 2.0 (1.296) | 0.9 (1.282)

3. Secondary Outcome: Mean Change From Baseline in Mean Flow Value in the Superotemporal Peripapillary Retina at Week 6
Description: Retinal perfusion assessments were made using Heidelberg Retinal Flowmetry (HRF). Assessments were made at 4 timepoints over a 12-hour period. Intensity of blood flow was measured in arbitrary units, with a higher number indicating an increased blood flow. An increase in ocular blood flow may reduce the risk of glaucoma progression.
Time Frame: Week 0, Week 6 (period-based)
Population: This reporting group includes all patients who received study medication and completed the on-therapy follow-up study visit in both periods (ITT). The analysis is based on patient eye-matched image data received.
Measure: Mean (Standard Error); unit: Arbitrary Units
Units Other Than Participants: eyes
Arm/Group | AZARGA | COMBIGAN
Number analyzed (Participants) | 32 | 32
Number analyzed (eyes) | 41 | 41
Arbitrary Units
  9:00 am | -272.4 (146.294) | -43.5 (146.586)
  1:00 pm | -12.1 (142.844) | 248.9 (144.917)
  5:00 pm | -26.7 (144.914) | -51.3 (142.844)
  9:00 pm | 14.0 (148.317) | -33.2 (144.451)

4. Secondary Outcome: Mean Change From Baseline in Mean Flow Value in the Inverotemporal Peripapillary Retina at Week 6
Description: as for outcome 3
Time Frame: Week 0, Week 6 (period-based)
Population: as for outcome 3
Measure: Mean (Standard Error); unit: Arbitrary Units
Units Other Than Participants: eyes
Arm/Group | AZARGA | COMBIGAN
Number analyzed (Participants) | 32 | 32
Number analyzed (eyes) | 41 | 41
Arbitrary Units
  9:00 am | 15.9 (92.064) | -70.0 (89.642)
  1:00 pm | -40.7 (89.642) | -89.2 (95.324)
  5:00 pm | -38.7 (88.363) | -69.1 (92.610)
  9:00 pm | 182.3 (92.064) | -91.0 (92.064)

5. Secondary Outcome: Mean Change From Baseline in Intraocular Pressure (IOP) at Week 6
Description: Intraocular pressure (IOP) is defined as the fluid pressure inside the eye. Intraocular pressure was measured with a calibrated pneumatonometer at 7 time points over a 24-hour period. High IOP (outside the normal range) can be a risk factor for developing glaucoma or glaucoma progression (leading to optic nerve damage).
Time Frame: Week 0, Week 6 (period-based)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: mmHg (millimeters of mercury)
Units Other Than Participants: eyes
Arm/Group | AZARGA | COMBIGAN
Number analyzed (Participants) | 32 | 32
Number analyzed (eyes) | 41 | 41
mmHg (millimeters of mercury)
  9:00 am | -6.3 (0.661) | -6.5 (0.661)
  1:00 pm | -6.0 (0.661) | -6.5 (0.661)
  5:00 pm | -5.6 (0.661) | -5.2 (0.661)
  9:00 pm | -4.3 (0.661) | -4.9 (0.661)
  12:00 am | -1.9 (0.661) | -1.6 (0.661)
  3:00 am | -1.3 (0.661) | -0.6 (0.661)
  6:00 am | -2.3 (0.668) | -1.2 (0.661)

6. Secondary Outcome: Mean Change From Baseline in Diastolic Blood Pressure at Week 6
Description: Blood pressure is defined as the pressure exerted by circulating blood upon the walls of the blood vessels, that is, arterial pressure of the systemic circulation of blood. Diastolic blood pressure refers to the minimum pressure, that is, the pressure between heartbeats. Diastolic glood pressure was measured at 7 timepoints in a 24-hour period using a calibrated sphygmomonometer. Higher blood pressure (outside the normal range) can be a risk factor for developing cardiovascular events, such as heart attack, stroke, or heart failure. Lower blood pressure (outside the normal range) can be a risk factor for dizziness or fainting.
Time Frame: Week 0, Week 6 (period-based)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: mmHg (millimeters of mercury)
Arm/Group | AZARGA | COMBIGAN
Number analyzed (Participants) | 32 | 32
mmHg (millimeters of mercury)
  9:00 am | -3.3 (1.315) | 0.6 (1.315)
  1:00 pm | -3.5 (1.315) | -4.3 (1.315)
  5:00 pm | -1.5 (1.315) | -0.9 (1.315)
  9:00 pm | -0.5 (1.315) | -2.1 (1.315)
  12:00 am | -1.4 (1.315) | -7.3 (1.315)
  3:00 am | -1.5 (1.315) | -3.8 (1.315)
  6:00 am | -0.5 (1.334) | -0.7 (1.315)

7. Secondary Outcome: Mean Change From Baseline in Systolic Blood Pressure at Week 6
Description: Blood pressure is defined as the pressure exerted by circulating blood upon the walls of the blood vessels, that is, arterial pressure of the systemic circulation of blood. Systolic blood pressure refers to the maximum pressure, that is, the pressure while the heart is beating, and was measured at 7 timepoints in a 24-hour period using a calibrated sphygmomonometer. Higher blood pressure (outside the normal range) can be a risk factor for developing cardiovascular events, such as heart attack, stroke, or heart failure. Lower blood pressure (outside the normal range) can be a risk factor for dizziness or fainting.
Time Frame: Week 0, Week 6 (period-based)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: mmHg (millimeters of mercury)
Arm/Group | AZARGA | COMBIGAN
Number analyzed (Participants) | 32 | 32
mmHg (millimeters of mercury)
  9:00 am | -4.2 (2.134) | 4.5 (2.134)
  1:00 pm | -2.6 (2.134) | -1.9 (2.134)
  5:00 pm | -2.9 (2.134) | -0.4 (2.134)
  9:00 pm | -1.4 (2.134) | -0.6 (2.134)
  12:00 am | -2.9 (2.134) | -12.2 (2.134)
  3:00 am | -2.9 (2.134) | -3.0 (2.134)
  6:00 am | -0.1 (2.165) | 3.0 (2.134)

8. Secondary Outcome: Mean Change From Baseline in Vascular Resistance in the Central Retinal Artery at Week 6
Description: Vascular resistance in the central retinal artery was assessed using Color Doppler Imaging (CDI). Assessments were made at 7 time points over a 24-hour period.
Time Frame: Week 0, Week 6 (period-based)
Population: as for outcome 3
Measure: Mean (Standard Error); unit: cm/s (centimeters per second)
Units Other Than Participants: eyes
Arm/Group | AZARGA | COMBIGAN
Number analyzed (Participants) | 32 | 32
Number analyzed (eyes) | 41 | 41
cm/s (centimeters per second)
  9:00 am | -0.00 (0.014) | 0.01 (0.014)
  1:00 pm | -0.01 (0.014) | 0.01 (0.014)
  5:00 pm | 0.00 (0.014) | -0.00 (0.014)
  9:00 pm | 0.00 (0.014) | 0.02 (0.014)
  12:00 am | 0.02 (0.014) | -0.01 (0.014)
  3:00 am | 0.01 (0.014) | 0.01 (0.014)
  6:00 am | -0.02 (0.014) | 0.02 (0.014)

9. Secondary Outcome: Mean Change From Baseline in Vascular Resistance in the Ophthalmic Artery at 6 Weeks
Description: Vascular resistance in the ophthalmic artery was assessed using Color Doppler Imaging (CDI). Assessments were made at 7 time points over a 24-hour period.
Time Frame: Week 0, Week 6 (period-based)
Population: as for outcome 3
Measure: Mean (Standard Error); unit: cm/s (centimeters per second)
Units Other Than Participants: eyes
Arm/Group | AZARGA | COMBIGAN
Number analyzed (Participants) | 32 | 32
Number analyzed (eyes) | 41 | 41
cm/s (centimeters per second)
  9:00 am | -0.01 (0.012) | -0.01 (0.011)
  1:00 pm | 0.02 (0.012) | 0.02 (0.012)
  5:00 pm | 0.01 (0.012) | 0.01 (0.012)
  9:00 pm | 0.01 (0.012) | 0.01 (0.011)
  12:00 am | -0.01 (0.012) | 0.02 (0.012)
  3:00 am | 0.01 (0.012) | 0.03 (0.012)
  6:00 am | 0.01 (0.012) | 0.03 (0.011)

10. Secondary Outcome: Mean Change From Baseline in End Diastolic Velocity in the Ophthalmic Artery at Week 6
Description: End diastolic velocity in the ophthalmic artery was assessed using Color Doppler Imaging (CDI). Assessments were made at 7 time points over a 24-hour period.
Time Frame: Week 0, Week 6 (period-based)
Population: as for outcome 3
Measure: Mean (Standard Error); unit: cm/s (centimeters per second)
Units Other Than Participants: eyes
Arm/Group | AZARGA | COMBIGAN
Number analyzed (Participants) | 32 | 32
Number analyzed (eyes) | 41 | 41
cm/s (centimeters per second)
  9:00 am | -0.0 (0.454) | -0.8 (0.448)
  1:00 pm | -0.6 (0.459) | -1.2 (0.460)
  5:00 pm | 0.5 (0.459) | 0.2 (0.466)
  9:00 pm | 0.4 (0.454) | -0.8 (0.448)
  12:00 am | -0.8 (0.466) | -1.4 (0.454)
  3:00 am | -0.1 (0.454) | -0.6 (0.459)
  6:00 am | -0.2 (0.466) | -0.5 (0.448)

11. Secondary Outcome: Mean Change From Baseline in Peak Systolic Velocity in the Ophthalmic Artery at Week 6
Description: Peak systolic velocity in the ophthalmic artery was assessed using Color Doppler Imaging (CDI). Assessments were made at 7 time points over a 24-hour period.
Time Frame: Week 0, Week 6 (period-based)
Population: as for outcome 3
Measure: Median (Standard Error); unit: cm/s (centimeters per second)
Units Other Than Participants: eyes
Arm/Group | AZARGA | COMBIGAN
Number analyzed (Participants) | 32 | 32
Number analyzed (eyes) | 41 | 41
cm/s (centimeters per second)
  9:00 am | -1.0 (1.237) | -3.8 (1.221)
  1:00 pm | -0.7 (1.251) | -1.4 (1.254)
  5:00 pm | 2.2 (1.251) | 1.3 (1.267)
  9:00 pm | 2.2 (1.237) | -1.4 (1.221)
  12:00 am | -2.3 (1.268) | -3.1 (1.235)
  3:00 am | 0.2 (1.235) | 0.0 (1.250)
  6:00 am | -0.6 (1.267) | 1.5 (1.221)

12. Secondary Outcome: Mean Change From Baseline in Peak Systolic Velocity in the Central Retinal Artery at Week 6
Description: Peak systolic velocity in the central retinal artery was assessed using Color Doppler Imaging (CDI). Assessments were made at 7 time points over a 24-hour period.
Time Frame: Week 0, Week 6 (period-based)
Population: as for outcome 3
Measure: Mean (Standard Error); unit: cm/s (centimeters per second)
Units Other Than Participants: eyes
Arm/Group | AZARGA | COMBIGAN
Number analyzed (Participants) | 32 | 32
Number analyzed (eyes) | 41 | 41
cm/s (centimeters per second)
  9:00 am | 0.9 (0.571) | 0.7 (0.565)
  1:00 pm | -0.2 (0.577) | 0.3 (0.578)
  5:00 pm | 1.0 (0.577) | 0.6 (0.565)
  9:00 pm | 0.9 (0.565) | -0.5 (0.565)
  12:00 am | 1.9 (0.577) | -0.5 (0.565)
  3:00 am | 0.2 (0.565) | -1.1 (0.570)
  6:00 am | 0.2 (0.571) | 0.9 (0.565)

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the duration of the study.
Description: The safety population is defined as patients who received study medication.
Arm/Group | AZARGA | COMBIGAN
Serious Adverse Events (participants affected / at risk) | 1/34 | 0/34
Other Adverse Events (participants affected / at risk) | 0/34 | 0/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AZARGA (N=34) | COMBIGAN (N=34)
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 — Recurrent Illness

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.